CLINICAL TRIAL: NCT01513395
Title: Focal Myometrial Contractions: Impact on Cervical Assessment and Association With Voiding. A Randomized Trial
Brief Title: Focal Myometrial Contractions: Impact on Cervical Assessment and Association With Voiding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, William Schnettler, Fellow in Maternal Fetal Medicine, Instructor, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2011-P-000425/2 BIDMC
Record Dates: First submitted 2012-01-17; First posted 2012-01-20 (Estimated); Last update posted 2012-01-23 (Estimated); Status verified 2012-01

CONDITIONS: Cervical Assessment; Focal Myometrial Contractions
Keywords: Cervical assessment; Focal myometrial contractions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate (No Intervention): Participants randomized to the "Immediate" or control arm (voiding within five minutes of cervical assessment), will undergo any indicated trans-abdominal ultrasound imaging and preparations for vaginal ultrasound (including readying the probe and preparing the exam table for lithotomy position) prior to using the restroom. The participant will be instructed to proceed to the restroom to empty her bladder completely. A synchronized clock will be placed in the restroom, and the patient will be asked to note the time that she completes voiding. This will be confirmed by the research staff by noting the time the participant enters and exits the restroom. Vaginal ultrasound and cervical assessment will then be performed immediately upon return to the ultrasound room (within a maximum of 5 minutes from voiding time).
- Interval (Experimental): Participants randomized to the "Interval" or experimental arm (cervical assessment 15 minutes or more after voiding) will be notified of their allocation and asked to immediately use the rest room and attempt to void completely. A synchronized clock will be located in this restroom, and each participant will be asked to note the time that she completes voiding. This will be confirmed by the research staff by noting the time the participant enters and exits the restroom. The participant will return to the waiting room or ultrasound room. Any indicated trans-abdominal ultrasound imaging will be performed, and preparations will be made for the vaginal ultrasound. The participant will be asked not to void prior to the vaginal ultrasound. Cervical assessment will take place at a minimum of 15 minutes from voiding time
  Interventions: Behavioral: Interval bladder emptying

INTERVENTIONS:
Behavioral: Interval bladder emptying — Participants randomized to the "Interval" arm (cervical assessment 15 minutes or more after voiding) will be notified of their allocation and asked to immediately use the rest room and attempt to void completely. A synchronized clock will be located in this restroom, and each participant will be asked to note the time that she completes voiding. This will be confirmed by the research staff by noting the time the participant enters and exits the restroom. The participant will return to the waiting room or ultrasound room. Any indicated trans-abdominal ultrasound imaging will be performed, and preparations will be made for the vaginal ultrasound. The participant will be asked not to void prior to the vaginal ultrasound. Cervical assessment will take place at a minimum of 15 minutes from voiding time.
  Arms: Interval

SUMMARY:
Focal myometrial (uterine) contractions occur in a substantial number of vaginal ultrasound examinations and can impede accurate cervical length measurement and placental location determination. The timing of bladder voiding is associated with the prevalence of focal myometrial contractions on vaginal ultrasound cervical assessment. We propose a blinded randomized-controlled trial of bladder voiding immediately before vaginal ultrasound for cervical assessment compared with no bladder voiding immediately before vaginal ultrasound in order to determine the prevalence of focal myometrial contractions during vaginal ultrasound cervical assessment and test whether timing of bladder voiding is associated with their incidence.

DETAILED DESCRIPTION:
This blinded randomized-controlled trial will be performed through the Division of Maternal Fetal Medicine at Beth Israel Deaconess Medical Center. We will offer enrollment to any pregnant woman at gestational weeks 14+0/7 through 31+6/7 presenting for obstetric ultrasound where cervical assessment and/or placental location determination is indicated. Patient positioning and image acquisition will follow a standard protocol and will be performed by the co-investigators. Outcome ascertainment will be performed by two co-investigators blinded to participant allocation upon completion of data collection. Demographic and obstetrical outcome data will be collected via review of the medical record. Analysis of primary and secondary outcomes will yield incidence data, and comparisons will be made between groups.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age of 14+0/7 through 31+6/7 weeks
* Presenting for obstetric ultrasound in the MFMU for cervical assessment and/or placental location determination
* Verbal consent
* Ability to refrain from urination for at least 15 minutes
* Age 18 years or greater

Exclusion Criteria:

* N/A

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-06 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Presence of focal myometrial contraction | Throughout the duration of that ultrasound examination (minutes)
  Focal myometrial contraction as defined by transvaginal ultrasound findings:
  * Thickening of the myometrial portion of the uterine wall visualized as two distinctly different areas of echogenicity
  * An unusually long-appearing cervix (possibly more than 50 mm) with an S-shaped endocervical canal and apparent internal os located appreciably cephalad
  * Asymmetric anterior and posterior lower uterine segment widths cephalad to apparent internal os
  * The thickening is transient.

SECONDARY OUTCOMES:
Location of focal myometrial contractions | Throughout the duration of that ultrasound examination (minutes)
  The location of focal myometrial contractions in relation to the internal cervical os is defined by:
  * Distance from internal os to caudal-most portion of focal myometrial contraction (measured with a curved line)..
  * Proportion that lie immediately adjacent to the internal cervical os.

CONTACTS AND LOCATIONS:
Overall Officials: Diana Rodriguez, MD, MPH, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- BIDMC - Dept. of Obstetrics and Gynecology, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Schnettler W, March M, Hacker MR, Modest AM, Rodriguez D. Impaired ultrasonographic cervical assessment after voiding: a randomized controlled trial. Obstet Gynecol. 2013 Apr;121(4):798-804. doi: 10.1097/AOG.0b013e3182860b8d. PMID 23635680